CLINICAL TRIAL: NCT00209703
Title: Feasibility Study of mFOLFOX6 (Oxaliplatin Combined With l-Leucovorin (l-LV) and 5-Fluorouracil) in Patients With Advanced Colorectal Cancer
Brief Title: Feasibility Study of mFOLFOX6 in Patients With Advanced Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Hokkaido Gastrointestinal Cancer Study Group (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGCSG0501
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-04-21 (Estimated); Status verified 2006-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Leucovorin; Fluorouracil

INTERVENTIONS:
Drug: Oxaliplatin
Drug: l-Leucovorin
Drug: 5-Fluorouracil

SUMMARY:
We performed a feasibility study of mFOLFOX6 in advanced colorectal cancer in Japan and to estimate the safety and efficacy of this regimen.

DETAILED DESCRIPTION:
A multicenter Open-label, single-arm feasibility study is conducted on patients with histological stage IV colorectal cancer given oxaliplatin, leucovorin plus fluorouracil. The usefulness of this regimens as therapy for colorectal cancer was evaluated by the disease-free survival rate (DFR), overall survival rate (OS), incidence and severity of adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of colorectral adenocarcinoma.
2. Measurable or assessable lesions.
3. Age: 15 ~ 75 years.
4. Performance Status (ECOG): 0 ~ 2.
5. Prior chemotherapy within 2 regimens.
6. Adequate function of major organs (bone marrow, heart, lungs, liver etc.). WBC 3,500/mm3. Hb 10.0 g/dl. Platelet count 100,000/mm3. GOT and GPT 2.5times the upper limit of normal (excluding liver metastasis). T-Bil 3.0mg/dl. Creatinine within the upper limit of normal. Normal ECG (not considering clinically unimportant arrhythmias and ischemic changes).

(10) Predicted survival for >8 weeks. (11) Able to give written informed consent.

Exclusion Criteria:

1. Severe pleural effusion or ascites.
2. Metastasis to the central nervous system (CNS).
3. Active gastrointestinal bleeding.
4. Active infection.
5. Uncontrolled ischemic heart disease.
6. Serious complications (such as intestinal paralysis, intestinal obstruction, interstitial pneumonia or pulmonary fibrosis, uncontrolled diabetes mellitus, heart failure, renal failure, or hepatic failure).
7. Active multiple cancer.
8. Severe mental disorder.
9. Pregnancy, possible pregnancy, or breast-feeding.
10. Patients with neuropathy ≥ grade 2
11. Judged to be ineligible for this protocol by the attending physician.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2005-01; Study Completion 2007-06

PRIMARY OUTCOMES:
Incidence and severity of adverse event

SECONDARY OUTCOMES:
Determine the clinical response rate, disease-free survival(DFS), overall survival(OS)

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Asaka, MD, PhD, Study Chair — Hokkaido Gastrointestinal Cancer Study Group
Locations (1):
- Hokkaido University Hospital (Hokkaido University Graduate School of Medicine), Sapporo, Hokkaido, Japan